CLINICAL TRIAL: NCT00673738
Title: Safety and Efficacy (Phase II) Study of Concurrent Cetuximab Plus Conformal Thoracic Radiotherapy in (Poor Prognosis) Patients With Inoperable or Unresectable, Locally Advanced Non-Small Cell Lung Cancer (LA - NSCLC)
Brief Title: Cetuximab Plus Conformal Thoracic Radiotherapy in Patients (Pts) With Inoperable or Unresectable Locally Advanced Non-Small Cell Lung Cancer (LA - NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15294; 106296 (Other: USF IRB); CA225286 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Results first posted 2014-03-04 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-09

CONDITIONS: Lung Cancer
Keywords: Lung; Thoracic; Immunotherapy; Radiotherapy; LA - NSCLC; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab; Docetaxel; Immunotherapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab Plus Radiotherapy (Experimental): Concurrent Cetuximab plus Conformal Thoracic Radiotherapy (CTRT). Patients were treated with definitive radiotherapy (70 Gy in 35 fractions, per our currently-existing institutional standard) with concurrent cetuximab followed by 3 cycles of consolidation docetaxel plus cetuximab.
  Interventions: Drug: Cetuximab; Radiation: Conformal Thoracic Radiotherapy (CTRT)

INTERVENTIONS:
Drug: Cetuximab — * Cetuximab dose: based on patient's actual weight. Loading phase dose of cetuximab is 400 mg/m2 IV administered over 120 minutes, on day 1 followed by; Concurrent phase, weekly infusion dose at 250 mg/m2 IV over 60 minutes, on days 8, 15, 22, 29, 36, 43, 50.
  * Radiation will be accompanied by weekly Cetuximab. Weekly Cetuximab will start on 1st day of radiation (Day 8). So, total number of cetuximab administrations will vary from 7 to 8. Patients will have every other week complete blood counts (CBCs), differentials, and blood urea nitrogen (BUN) plus creatinine and Mg. If patient's ANC drops below 1,000 and/or the platelet count below 75,000 during CTRT, the corresponding, weekly dose of cetuximab will be omitted.
  Other Names: Chemotherapy single agent systemic; docetaxel; immunotherapy
Radiation: Conformal Thoracic Radiotherapy (CTRT) — * Radiation will be accompanied by weekly Cetuximab. Weekly Cetuximab will start on 1st day of radiation (Day 8). So, total number of cetuximab administrations will vary from 7 to 8. Patients will have every other week CBCs, differentials, and BUN plus creatinine and Mg. If patient's ANC drops below 1,000 and/or the platelet count below 75,000 during CTRT, the corresponding, weekly dose of cetuximab will be omitted.
  * Radiation therapy will begin on day 8 (with window of ± 3 days). Adequate hematologic profile (ANC >1,000 and platelets >75,000) required. Patient may be delayed for a max. of 2 weeks. If > 2 week delay occurs, patient will come off study.
  Other Names: CTRT; Radiotherapy

SUMMARY:
This research is being done to find out if a treatment consisting of a combination of thoracic radiotherapy with cetuximab, given together, and followed by chemotherapy with docetaxel and cetuximab (also given together) will kill the cancer cells in the patient's body and shrink the size of their tumor without causing unacceptable side effects. This may allow patients to live longer or decrease the frequency and/or severity of the symptoms caused by the cancer without increasing the frequency and/or severity of the symptoms caused by the treatment.

DETAILED DESCRIPTION:
Patients will be asked to spend about six months in this study. There will be 4 different phases in this study as follows: (1) Loading Phase: This is the first week (week 1) of the study, when patients receive their first (loading) dose of cetuximab only, in the vein. (2) Concurrent Phase: During this phase patients will be treated simultaneously (concurrently) with radiation therapy to their chest and cetuximab. Radiation is delivered 5 days a week, Monday to Friday for a total of 7 weeks (weeks 2-8). Cetuximab is delivered in the vein, weekly, during the weeks of radiation. (3) Recovery Phase: Patients receive no treatment during these next 3 weeks (weeks 9-11). This phase is designed to allow patients to recover from side effects before they start the last phase. (4) Consolidation Phase: The last phase. Patients will receive 3 doses of chemotherapy with docetaxel during this phase. Docetaxel is given intravenously every 21 days. Patients also receive weekly cetuximab during this phase. Cetuximab is delivered in a similar way as it was during the concurrent (second) phase of this study. In total, this phase lasts 6 weeks (weeks 12-18). Once the therapy treatment is completed, and if the patient's cancer did not get worse, follow up visits will include visits to their physician every three months for 2 years, then every 4 months for 2 years or more, as long as their cancer doesn't get worse (at which time they will be removed from the study).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed inoperable or unresectable, LA-NSCLC (adenocarcinoma, squamous cell carcinoma or anaplastic large cell carcinoma or non-small cell otherwise not specified).
* Eligible Stages: Stages IIA through IIIA disease if it is felt that they are not candidates for possible resection, medically or otherwise. Stage IIIA (multi-station mediastinal lymph nodes) and stage IIIB disease without significant pleural effusion (metastases to contralateral mediastinal or supraclavicular lymph nodes) are also eligible.
* Age ≥ 70 OR Eastern Cooperative Oncology Group (ECOG) performance status (PS) = 2 at time of registration OR weight loss ≥ 5% in the preceding three months to the time of registration
* Must have measurable disease by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. When applicable, baseline measurements/evaluations must be obtained within 4 weeks prior to registration.
* Must have adequate bone marrow reserve as determined by the following laboratory values, obtained within 14 days prior to registration:

  * White blood cell count (WBC) ≥ 4000/ul or absolute neutrophil count (ANC) ≥ 1000/ul
  * Platelet count ≥ 100,000/ul
  * Hemoglobin ≥ 8 gms/dl
* Adequate renal and liver function as determined by the following laboratory values, obtained within 14 days prior to registration:

  * Serum creatinine ≤ 2.0 mg/dl or creatinine clearance ≥ 40 cc/min
  * Bilirubin < 2.0 mg/dl
  * serum glutamic oxaloacetic transaminase (SGOT) ≤ 2.5 times the upper limit of normal(ULN)
* Written, informed consent must be obtained prior to registration
* Women of childbearing potential (WOCBP) must use an accepted, effective method of contraception during the course of the study, in a manner such that risk of failure is minimized. Sexually active males enrolled should understand the risks to any sexual partner of childbearing potential; must also practice an effective method of contraception. WOCBP must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy; have a negative pregnancy test within 7 days prior to first receiving investigational product; be instructed to contact the Investigator immediately if they suspect they might be pregnant at any time during study participation. Investigator must immediately notify Bristol-Myers Squibb (BMS) in the event of a confirmed pregnancy in a patient participating in the study. If the pregnancy test is positive, the patient must not receive investigational product and must not be enrolled in the study.

Exclusion Criteria:

* Must not have small cell carcinoma as part of the histological specimen
* Evidence of distant metastasis.
* History of a prior or concomitant malignancy in the past 3 years except for surgically cured basal cell carcinoma of the skin or carcinoma in situ of the cervix. Invasive malignancies, properly treated and currently disease-free > 3 years are allowed.
* Prior thoracic radiotherapy or epidermal growth factor receptor (EGFR) pathway targeting therapy. Prior systemic chemotherapy is allowed if received as therapy for an invasive malignancy, currently disease-free > 3 years
* Concomitant life threatening or uncontrolled serious medical illness such as cardiac disease (uncontrolled hypertension, arrhythmia, unstable angina, recent myocardial infarction, end stage congestive heart failure, cardiomyopathy with decreased ejection fraction), liver disease with significant hepatic insufficiency, kidney disease with significant renal insufficiency or organic brain syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-04; Primary Completion 2013-12 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Chiappori, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Moffitt Cancer Center from May, 2008 to November, 2010.
Groups:
- Cetuximab Plus Radiotherapy: Concurrent Cetuximab plus Conformal Thoracic Radiotherapy (CTRT)
Period: Overall Study
Arm/Group | Cetuximab Plus Radiotherapy
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cetuximab Plus Radiotherapy
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 25
Age, Continuous [Median (Full Range); unit: years] | 72 [58 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival (PFS)
Description: Progression Free Survival is defined as the interval between the date of the first cetuximab administration and the date of objective progression of disease. Progression was evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST) Criteria. Progressive Disease (PD): Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Up to 36 months
Population: All participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus Radiotherapy
Number analyzed (Participants) | 27
months | 7.5 [4.0 to 10.7]

2. Secondary Outcome: Median Overall Survival (OS)
Description: Overall survival is defined as the time from randomization until death from any cause.
Time Frame: Up to 36 months
Population: All participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus Radiotherapy
Number analyzed (Participants) | 27
months | 10.5 [4.3 to 20.5]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR = Complete Response (CR) + Partial Response (CR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.0. Complete Response: Disappearance of all target lesions; Partial Response: At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: Up to 36 months
Population: All participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab Plus Radiotherapy
Number analyzed (Participants) | 27
percentage of participants
  Partial Response | 59.3 [38.8 to 77.6]
  Complete Response | 0 [NA to NA] — There was no occurrence of Complete Response.

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Cetuximab Plus Radiotherapy
Serious Adverse Events (participants affected / at risk) | 20/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab Plus Radiotherapy (N=27)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1
Low Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2
Supraventricular and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 2
Sweating (diaphoresis) (General disorders) | 1
Death not associated with CTCAE term - Death (General disorders) | 2
Death not associated with CTCAE term - Sudden death (General disorders) | 2
Anorexia (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 1
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 3
Esophagitis (Gastrointestinal disorders) | 2
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Stricture/stenosis (including anastomotic), GI - Esophagus (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Hemorrhage, pulmonary/upper respiratory - Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 1
Febrile neutropenia (Infections and infestations) | 4
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Lung (Infections and infestations) | 1
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Urinary Tract (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Esophagus (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 4
Infection with normal ANC or Grade 1 or 2 neutrophils - Skin (cellulitis) (Infections and infestations) | 1
Edema: limb (Blood and lymphatic system disorders) | 1
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 1
Mood alteration - Agitation (General disorders) | 1
Pain - Abdomen NOS (General disorders) | 1
Pain - Throat/pharynx/larynx (General disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab Plus Radiotherapy (N=27)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 19
Esophagitis (Gastrointestinal disorders) | 19
Constipation (Gastrointestinal disorders) | 15
Nausea (Gastrointestinal disorders) | 14
Anorexia (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 6
Dehydration (Gastrointestinal disorders) | 5
Stricture/stenosis (including anastomotic), GI - Esophagus (Gastrointestinal disorders) | 4
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 4
Heartburn/dyspepsia (Gastrointestinal disorders) | 2
Mucositis/stomatitis clinical exam) - Oral cavity (Gastrointestinal disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 22
Weight loss (General disorders) | 5
Constitutional Symptoms - Other (General disorders) | 4
Insomnia (General disorders) | 4
Fever (in the absence of neutropenia) (Infections and infestations) | 2
Sweating (diaphoresis) (General disorders) | 2
Rash: dermatitis associated with radiation - Radiation (Skin and subcutaneous tissue disorders) | 20
Pruritus/itching (Skin and subcutaneous tissue disorders) | 19
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 18
Dry skin (Skin and subcutaneous tissue disorders) | 9
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 5
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Nail changes (Skin and subcutaneous tissue disorders) | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 2
Pain - Head/headache (General disorders) | 6
Pain - Back (General disorders) | 4
Pain - Chest/thorax NOS (General disorders) | 4
Pain - Throat/pharynx/larynx (General disorders) | 4
Pain - Abdomen NOS (General disorders) | 3
Pain - Esophagus (General disorders) | 2
Pain - Other (General disorders) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 4
Febrile neutropenia (fever of unknown origin) (Infections and infestations) | 3
Infection with normal ANC or Grade 1 or 2 neutrophils - Bronchus (Infections and infestations) | 2
Infection with unknown ANC - Oral cavity-gums (gingivitis) (Infections and infestations) | 2
Dizziness (General disorders) | 6
Confusion (General disorders) | 2
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 5
Muscle weakness generalized or specific area (not due to neuropathy) whole body/generalized (Musculoskeletal and connective tissue disorders) | 4
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 4
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2
Edema: limb (Blood and lymphatic system disorders) | 4
Edema: head and neck (Blood and lymphatic system disorders) | 2
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 4
Hypotension (Cardiac disorders) | 4
Ocular/Visual - Other (Eye disorders) | 2
Thrombosis/thrombus/embolism (Vascular disorders) | 2
Low Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2

LIMITATIONS AND CAVEATS:
Accrual, and therefore treatment ended earlier than planned due to pulmonary toxicity. Three participants remain on follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes